CLINICAL TRIAL: NCT02418000
Title: A Phase 1/2a Study of E6201 for the Treatment of Advanced Hematologic Malignancies With FLT3 and/or Ras Mutations, Including Acute Myeloid Leukemia (AML), Myelodysplastic Syndrome (MDS) or Chronic Myelomonocytic Leukemia (CMML)
Brief Title: A Study of E6201 for the Treatment of Advanced Hematologic Malignancies With FLT3 and/or Ras Mutations
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Insufficient efficacy in Phase 1 dose-escalation portion of study
Sponsor: Spirita Oncology, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BSC-101-01
Record Dates: First submitted 2015-02-18; First posted 2015-04-16 (Estimated); Results first posted 2019-03-05 (Actual); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: AML; MDS; CMML
MeSH Terms: interventions — 14-(ethylamino)-8,9,16-trihydroxy-3,4-dimethyl-3,4,9,19-tetrahydro-1H-2-benzoxacyclotetradecine-1,7(8H)-dione

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- E6201 240 mg/m^2 IV weekly (Experimental): E6201 240 mg/m^2 administered IV over 2 hours once weekly, on Days 1, 8, 15, and 22, repeated every 28 days (= 1 cycle)
  Interventions: Drug: E6201
- E6201 320 mg/m^2 IV weekly (Experimental): E6201 320 mg/m^2 administered IV over 2 hours once weekly, on Days 1, 8, 15, and 22, repeated every 28 days (= 1 cycle)
  Interventions: Drug: E6201
- E6201 160 mg/m^2 IV twice weekly (Experimental): E6201 160 mg/m^2 administered IV over 2 hours twice weekly, on Days 1, 4, 8, 11, 15, 18, 22 and 25, repeated every 28 days (= 1 cycle)
  Interventions: Drug: E6201
- E6201 240 mg/m^2 IV twice weekly (Experimental): E6201 240 mg/m^2 administered IV over 2 hours twice weekly, on Days 1, 4, 8, 11, 15, 18, 22 and 25, repeated every 28 days (= 1 cycle)
  Interventions: Drug: E6201
- E6201 320 mg/m^2 IV twice weekly (Experimental): E6201 320 mg/m^2 administered IV over 2 hours twice weekly, on Days 1, 4, 8, 11, 15, 18, 22, and 25, repeated every 28 days (= 1 cycle)
  Interventions: Drug: E6201

INTERVENTIONS:
Drug: E6201 — Single Group Assignment
  Other Names: Dual inhibitor of FLT3 and MEK1

SUMMARY:
This is a Phase 1/2a dose-escalation study of E6201, a dual mitogen-activated protein kinase/extracellular-signal regulated kinase 1 (MEK1) and FMS-like tyrosine kinase 3 (FLT3) inhibitor, in subjects with advanced hematologic malignancies with documented FLT3 and/or rat sarcoma (Ras) mutations. The Phase1 portion of the study will be a safety run-in (up to 30 subjects) to establish a recommended Phase 2 dose (RP2D). The Ph. 2a portion of the study will evaluate three specific patients groups: Cohort 1 will enroll patients with relapsed or refractory AML and confirmed FLT3 mutation (with or without a Ras mutation) without prior exposure to a FLT3 inhibitor; Cohort 2 will enroll patients with relapsed or refractory AML and confirmed FLT3 mutation (with or without a Ras mutation) with prior exposure to a FLT3 inhibitor; Cohort 3 will enroll patients with relapsed or refractory AML with a confirmed Ras mutation and no FLT3 mutation.

DETAILED DESCRIPTION:
Phase 1 (Safety Run-In): Following Screening, a total of up to 30 subjects in up to 5 dose cohorts to establish the RP2D. The safety run-in phase will be a standard 3+3 cohort design.

Phase 2a (Expansion): Once the Phase 1 Safety Run-In portion of the study is complete and an RP2D is established, additional subjects will be enrolled into the Phase 2 Expansion portion in three cohorts. Cohort 1 will enroll up to 26 patients with relapsed or refractory AML and confirmed FLT3 mutation (with or without a Ras mutation) without prior exposure to a FLT3 inhibitor. Cohort 2 will enroll up to 26 patients with relapsed or refractory AML and confirmed FLT3 mutation (with or without a Ras mutation) with prior exposure to a FLT3 inhibitor. Cohort 3 will enroll up to 10 patients with relapsed or refractory AML with a confirmed Ras mutation and no FLT3 mutation. Cohort 1 and 2 of the Expansion Phase will incorporate a Simon 2-stage optimal design. Subjects with AML enrolled in the Phase 1 portion of the study at the RP2D will count towards the Phase 2a accrual for the appropriate cohort.

Subjects will receive E6201 weekly or bi-weekly on a 28-day schedule, with the schedule and dose level established in the Safety Run-In portion of the study. Disease assessments, including analysis of blood and bone marrow samples, will be performed at the end of Cycles 1 and 3 and every 2 cycles thereafter. Disease assessments may be made at other time points at the discretion of the Investigator.

Subjects who demonstrate clinical benefit (objective response or stable disease) will be allowed to continue therapy with E6201 until progression of disease, observation of unacceptable adverse events, intercurrent illness or changes in the patient's condition that prevents further study participation.

During the study, ECGs will be performed, blood will be collected for hematology, serum chemistry, pharmacokinetics and pharmacodynamics assessments, and bone marrow will be collected for the assessment of disease response and mutational status.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ≥ 18 years of age
* Phase 1: Confirmed relapsed or refractory AML with a documented FLT3 and/or Ras mutation, or ≥ 60 years with newly diagnosed FLT3+ and/or Ras+ AML and not eligible for standard induction chemotherapy or FLT3+ and/or Ras+ higher-risk MDS/CMML (defined as ≥ 10% marrow blasts or ≥ 5% peripheral blood blasts or Revised International Prognostic Scoring System [IPSS-R] score ≥ 3.5) and relapsed or refractory to prior therapy
* Phase 2: Confirmed relapsed or refractory AML with a documented FLT3 and/or Ras mutation, or age ≥ 60 years with newly diagnosed FLT3+ and/or Ras+ AML and not eligible for standard induction chemotherapy
* At least 3 weeks beyond the last cancer treatment for the disease under study, major surgery and recovered from all acute toxicities (≤ Grade 1) by first dose of study drug (C1D1). Hydroxyurea used to control peripheral blast counts is permitted during the first 2 cycles.
* Adequate performance status Eastern Cooperative Oncology Group (ECOG) ≤ 2
* Adequate renal and hepatic function:

  * creatinine ≤ 1.5 mg/dL OR calculated creatinine clearance ≥ 45 mL/minute
  * total bilirubin ≤ 2 times the upper limit of normal (ULN) unless due to Gilbert's disease or thought to be due to underlying AML
  * ALT and AST ≤ 5 times ULN
* Negative serum pregnancy test within 14 days prior to the first dose of study therapy for women of child-bearing potential (WCBP). Sexually active WCBP and male subjects must agree to use adequate methods to avoid pregnancy throughout the study and for 28 days after completion of study treatment.
* Ability to provide written informed consent

Exclusion Criteria:

* History of clinically significant cardiac impairment, congestive heart failure (CHF) New York Heart Association (NYHA) Class III or IV, unstable angina, or myocardial infarction during the previous 6 months, or serious cardiac arrhythmia
* QT interval corrected for rate (QTc) ≥ 450 msec for males and ≥ 460 msec for females on the ECG obtained at Screening using Fridericia method for QTc calculation (average of 3 readings)
* Concomitant medication(s) that may cause QTc prolongation or induce Torsades de Pointes with the exception of anti-microbials used as standard of care to prevent or treat infections and other such drugs that are considered by the investigator to be essential for the care of the patient. However, if such medications are deemed to be necessary during the study, more extensive ECG monitoring will be added during the period of concomitant drug administration.
* Presence of active central nervous system (CNS) leukemia. Subjects adequately treated for CNS leukemia documented by 2 consecutive cerebrospinal fluid samples negative for leukemia cells are eligible. Subjects with no history of CNS leukemia will not be required to undergo cerebrospinal fluid sampling for eligibility.
* Known positive for human immunodeficiency virus (HIV), hepatitis B virus surface antigen (HBsAg), or hepatitis C virus HCV)
* Active, uncontrolled infection
* Known hypersensitivity to any study drug component
* History of another malignancy; Exception: Patients disease-free for 2 years or treated in situ carcinoma
* Any other medical intervention or other condition which, in the opinion of the Principal Investigator, could compromise adherence to study requirements or confound the interpretation of study results
* Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2015-04-10; Primary Completion 2017-06-08 (Actual); Study Completion 2017-06-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gautam Borthakur, MD, Study Chair — MD Anderson Cancer Center Houston, TX 77030
Locations (4):
- United States (4):
  - Colorado Blood Cancer Institute, Denver, Colorado
  - H. Lee Moffitt Cancer Center & research Institute, Tampa, Florida
  - MD Anderson Cancer Center, Houston, Texas
  - Texas Transplant Institute, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Responsible Party URL — http://www.StrategiaTx.com

RESULTS

PARTICIPANT FLOW:
Groups:
- E6201 240 mg/m^2 Weekly: Cohort 1: Participants were administered E6201 240 mg/m^2 IV over 2 hours once weekly, on Days 1, 8, 15, and 22, repeated every 28 days (= 1 cycle) until progression of disease, toxicity or other reason for discontinuation of study drug, and followed for up to 6 months after the last dose.
- E6201 320 mg/m^2 Weekly: Cohort 2: Participants were administered E6201 320 mg/m^2 IV over 2 hours once weekly, on Days 1, 8, 15, and 22, repeated every 28 days (= 1 cycle) until progression of disease, toxicity or other reason for discontinuation of study drug, and followed for up to 6 months after the last dose.
- E6201 160 mg/m^2 Twice Weekly: Cohort 3: Participants were administered E6201 160 mg/m^2 IV over 2 hours twice weekly, on Days 1, 4, 8, 11, 15, 18, 22 and 25, repeated every 28 days (= 1 cycle) until progression of disease, toxicity or other reason for discontinuation of study drug, and followed for up to 6 months after the last dose.
- E6201 240 mg/m^2 Twice Weekly: Cohort 4: Participants were administered E6201 240 mg/m^2 IV over 2 hours twice weekly, on Days 1, 4, 8, 11, 15, 18, 22 and 25, repeated every 28 days (= 1 cycle) until progression of disease, toxicity or other reason for discontinuation of study drug, and followed for up to 6 months after the last dose.
- E6201 320 mg/m^2 Twice Weekly: Cohort 5: Participants were administered E6201 320 mg/m^2 IV over 2 hours twice weekly, on Days 1, 4, 8, 11, 15, 18, 22 and 25, repeated every 28 days (= 1 cycle) until progression of disease, toxicity or other reason for discontinuation of study drug, and followed for up to 6 months after the last dose.
Period: Cohort 1: E6201 240 mg/m^2 Weekly
Arm/Group | E6201 240 mg/m^2 Weekly | E6201 320 mg/m^2 Weekly | E6201 160 mg/m^2 Twice Weekly | E6201 240 mg/m^2 Twice Weekly | E6201 320 mg/m^2 Twice Weekly
Started | 7 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 7 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 4 | 0 | 0 | 0 | 0
Not completed — Prepare for HSCT | 1 | 0 | 0 | 0 | 0
Period: Cohort 2: E6201 320 mg/m^2 Weekly
Arm/Group | E6201 240 mg/m^2 Weekly | E6201 320 mg/m^2 Weekly | E6201 160 mg/m^2 Twice Weekly | E6201 240 mg/m^2 Twice Weekly | E6201 320 mg/m^2 Twice Weekly
Started | 0 | 10 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 10 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 9 | 0 | 0 | 0
Period: Cohort 3: 160 mg/m^2 Twice Weekly
Arm/Group | E6201 240 mg/m^2 Weekly | E6201 320 mg/m^2 Weekly | E6201 160 mg/m^2 Twice Weekly | E6201 240 mg/m^2 Twice Weekly | E6201 320 mg/m^2 Twice Weekly
Started | 0 | 0 | 3 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 3 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 3 | 0 | 0
Period: Cohort 4: 240 mg/m^2 Twice Weekly
Arm/Group | E6201 240 mg/m^2 Weekly | E6201 320 mg/m^2 Weekly | E6201 160 mg/m^2 Twice Weekly | E6201 240 mg/m^2 Twice Weekly | E6201 320 mg/m^2 Twice Weekly
Started | 0 | 0 | 0 | 3 | 0
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 3 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 3 | 0
Period: Cohort 5: 320 mg/m^2 Twice Weekly
Arm/Group | E6201 240 mg/m^2 Weekly | E6201 320 mg/m^2 Weekly | E6201 160 mg/m^2 Twice Weekly | E6201 240 mg/m^2 Twice Weekly | E6201 320 mg/m^2 Twice Weekly
Started | 0 | 0 | 0 | 0 | 4
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 4
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1: E6201 240 mg/m^2 Weekly: Cohort 1: Participants were administered E6201 240 mg/m^2 IV over 2 hours once weekly, on Days 1, 8, 15, and 22, repeated every 28 days (= 1 cycle) until progression of disease, toxicity or other reason for study drug discontinued, and followed for up to 6 months after the last dose.
- Cohort 2: E6201 320 mg/m^2 Weekly: Cohort 2: Participants were administered E6201 320 mg/m^2 IV over 2 hours once weekly, on Days 1, 8, 15, and 22, repeated every 28 days (= 1 cycle) until progression of disease, toxicity or other reason for study drug discontinuation, and followed for up to 6 months after the last dose.
- Cohort 3: E6201 160 mg/m^2 Twice Weekly: Cohort 3: Participants were administered E6201 160 mg/m^2 IV over 2 hours twice weekly, on Days 1, 4, 8, 11, 15, 18, 22 and 25, repeated every 28 days (= 1 cycle) until progression of disease, toxicity or other reason for study drug discontinuation, and followed for up to 6 months after the last dose.
- Cohort 4: E6201 240 mg/m^2 Twice Weekly: Cohort 4: Participants were administered E6201 240 mg/m^2 IV over 2 hours twice weekly, on Days 1, 4, 8, 11, 15, 18, 22 and 25, repeated every 28 days (= 1 cycle) until progression of disease, toxicity or other reason for study drug discontinuation, and followed for up to 6 months after the last dose.
- Cohort 5: E6201 320 mg/m^2 Twice Weekly: Cohort 5: Participants were administered E6201 320 mg/m^2 IV over 2 hours twice weekly, on Days 1, 4, 8, 11, 15, 18, 22 and 25, repeated every 28 days (= 1 cycle) until progression of disease, toxicity or other reason for study drug discontinuation, and followed for up to 6 months after the last dose.
- Total: Total of all reporting groups
Arm/Group | Cohort 1: E6201 240 mg/m^2 Weekly | Cohort 2: E6201 320 mg/m^2 Weekly | Cohort 3: E6201 160 mg/m^2 Twice Weekly | Cohort 4: E6201 240 mg/m^2 Twice Weekly | Cohort 5: E6201 320 mg/m^2 Twice Weekly | Total
Number analyzed (Participants) | 7 | 10 | 3 | 3 | 4 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.57 (13.97) | 51.10 (19.14) | 61.33 (11.02) | 56.33 (12.01) | 56.00 (17.64) | 56.26 (15.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 2 | 1 | 2 | 14
  Male | 2 | 6 | 1 | 2 | 2 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 1 | 0 | 0 | 3
  Not Hispanic or Latino | 4 | 8 | 2 | 3 | 4 | 21
  Unknown or Not Reported | 2 | 1 | 0 | 0 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 3 | 0 | 0 | 0 | 4
  White | 5 | 6 | 3 | 2 | 3 | 19
  More than one race | 1 | 1 | 0 | 0 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 10 | 3 | 3 | 4 | 27
Disease Type [Count of Participants; unit: Participants]
  AML | 4 | 10 | 3 | 3 | 4 | 24
  MDS | 1 | 0 | 0 | 0 | 0 | 1
  CMML | 2 | 0 | 0 | 0 | 0 | 2
Eastern Cooperative Group (ECOG) Performance Status [Count of Participants; unit: Participants] — ECOG Performance Status:
  0 = Fully active, able to carry on all pre-disease performance without restriction
  1. = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  2. = Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours
  3. = Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours
  4. = Completely disabled. Cannot carry on any selfcare. Totally confined to bed or chair
  5. = Dead
  Participants
    0 | 2 | 1 | 0 | 0 | 0 | 3
    1 | 5 | 6 | 2 | 3 | 4 | 20
    2 | 0 | 3 | 1 | 0 | 0 | 4
    3 | 0 | 0 | 0 | 0 | 0 | 0
    4 | 0 | 0 | 0 | 0 | 0 | 0
Prior Cancer Therapies [Median (Full Range); unit: Number of treatment regimens]
  All Prior Cancer Treatment Regimens | 3 [2 to 8] | 6.5 [4 to 14] | 4 [4 to 7] | 5 [4 to 10] | 4 [4 to 11] | 5 [2 to 14]
  Prior FLT3 Inhibitor Treatment Regimens | 1 [1 to 1] | 1 [1 to 3] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 3]

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of E6201
Description: Phase 1 (Safety Run-In) was conducted in 5 dose cohorts in up to 30 subjects in a standard 3+3 dose-escalation design to establish an MTD and recommended Phase 2 dose (RP2D). Safety assessed through the monitoring of adverse events (AEs), serious adverse events (SAEs), clinical laboratory parameters (hematology and serum chemistry), vital sign measurements, electrocardiograms (ECGs) and physical examinations.
Time Frame: Up to 6 weeks for each dose cohort
Population: Full analysis set (FAS): All subjects who were administered any fraction of a dose of study medication
Measure: Number; unit: E6201 MTD (mg/m^2) IV twice weekly
Groups:
- All Participants: All study participants who received at least 1 dose of E6201 at 240 or 320 mg/m^2 IV weekly, or at 160, 240 or 320 mg/m^2 IV twice weekly
Arm/Group | All Participants
Number analyzed (Participants) | 27
E6201 MTD (mg/m^2) IV twice weekly | 320

2. Primary Outcome: Number of Participants Who Experienced Dose-Limiting Toxicities (DLTs)
Description: A DLT was defined as any one of the following events: prolonged myelosuppression (as defined by the National Cancer Institute [NCI] criteria specific for leukemia, i.e., marrow cellularity < 5% at ≥ 6 weeks from start of therapy without evidence of leukemia); ≥ Grade 3 non-hematologic toxicity (excluding Grade 3 nausea, vomiting or diarrhea that is adequately controlled with supportive care and resolves to ≤ Grade 2 within 48 hours, or Grade 3 electrolyte disturbances responsive to correction within 24 hours); ≥ Grade 3 liver function tests (LFTs) lasting > 7 days; treatment interruption > 14 days due to toxicity; or other important medical event.
  DLTs were collected to determine the MTD which is defined as the dose level below the dose at which ≥ 2 of 6 patients in a dose cohort experienced a DLT.
Time Frame: Up to 6 weeks for each dose cohort
Population: Full analysis set (FAS): All subjects who were administered any fraction of a dose of study medication.
Measure: Number; unit: Number of Participants with DLTs
Groups:
- E6201 240 mg/m^2 Weekly: E6201 240 mg/m^2 IV over 2 hours once weekly, on Days 1, 8, 15, and 22, repeated every 28 days (= 1 cycle) until progression of disease, toxicity or other reason for discontinuation of study drug, and followed for up to 6 months after the last dose.
- E6201 320 mg/m^2 Weekly: E6201 320 mg/m^2 IV over 2 hours once weekly, on Days 1, 8, 15, and 22, repeated every 28 days (= 1 cycle) until progression of disease, toxicity or other reason for discontinuation of study drug, and followed for up to 6 months after the last dose.
- E6201 160 mg/m^2 Twice Weekly: E6201 160 mg/m^2 IV over 2 hours twice weekly, on Days 1, 4, 8, 11, 15, 18, 22 and 25, repeated every 28 days (= 1 cycle) until progression of disease, toxicity or other reason for discontinuation of study drug, and followed for up to 6 months after the last dose.
- E6201 240 mg/m^2 Twice Weekly: E6201 240 mg/m^2 IV over 2 hours twice weekly, on Days 1, 4, 8, 11, 15, 18, 22 and 25, repeated every 28 days (= 1 cycle) until progression of disease, toxicity or other reason for discontinuation of study drug, and followed for up to 6 months after the last dose.
- E6201 320 mg/m^2 IV Twice Weekly: E6201 320 mg/m^2 IV over 2 hours twice weekly, on Days 1, 4, 8, 11, 15, 18, 22 and 25, repeated every 28 days (= 1 cycle) until progression of disease, toxicity or other reason for discontinuation of study drug, and followed for up to 6 months after the last dose.
Arm/Group | E6201 240 mg/m^2 Weekly | E6201 320 mg/m^2 Weekly | E6201 160 mg/m^2 Twice Weekly | E6201 240 mg/m^2 Twice Weekly | E6201 320 mg/m^2 IV Twice Weekly
Number analyzed (Participants) | 7 | 10 | 3 | 3 | 4
Number of Participants with DLTs | 1 | 1 | 0 | 0 | 0

3. Secondary Outcome: Overall Response Rate
Description: For acute myeloid leukemia (AML): Revised Recommendations of the International Working Group (IWG) Response Criteria for AML: CR: Free of leukemia-related symptoms, absolute neutrophil count (ANC) > 1.0 x 10^9/L, platelet count ≥ 100 x 10^9/L, normal bone marrow with < 5% blasts and no Auer rods. CRi: As per CR but w/ residual thrombocytopenia (platelet count <100 x 10^9/L) or residual neutropenia (ANC <1.0 x 10^9/L). PR: ≥50% decrease bone marrow blasts to 5 - 25% abnormal cells, or CR w/ ≤ 5% blasts if Auer rods present.
  For myelodysplastic syndrome (MDS) and chronic myelomonocytic leukemia (CMML): Modified IWG Response Criteria for MDS: CR: Free of leukemia-related symptoms, ANC ≥1.0 x 10^9/L, platelet count ≥100 x 10^9/L, bone marrow ≤5% myeloblasts, normal maturation of all cell lines, hemoglobin ≥ 11g/dL, no blasts in the peripheral blood. PR: All CR criteria w/ ≥50% decrease in bone marrow blasts over pre-treatment, but still > 5%.
Time Frame: At the end of C1 and every 2 cycles thereafter through 6 months following last dose of study drug
Population: The analysis population was the per-protocol set (PPS). The PPS included all subjects in the FAS who had a valid baseline and one or more post-treatment assessments for a specified measure.
Measure: Number; unit: Objective Responses
Groups:
- E6201 320 mg/m^2 Twice Weekly: E6201 320 mg/m^2 IV over 2 hours twice weekly, on Days 1, 4, 8, 11, 15, 18, 22 and 25, repeated every 28 days (= 1 cycle) until progression of disease, toxicity or other reason for discontinuation of study drug, and followed for up to 6 months after the last dose.
Arm/Group | E6201 240 mg/m^2 Weekly | E6201 320 mg/m^2 Weekly | E6201 160 mg/m^2 Twice Weekly | E6201 240 mg/m^2 Twice Weekly | E6201 320 mg/m^2 Twice Weekly
Number analyzed (Participants) | 7 | 10 | 3 | 3 | 4
Objective Responses | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Duration of Response
Description: Length of time from the first evidence of objective response to the first evidence of progression
Time Frame: At the end of C1 and every 2 cycles thereafter through 6 months following last dose of study drug
Population: The analysis population was the per-protocol set (PPS). The PPS included all subjects in the FAS who had a valid baseline and one or more post-treatment assessments for a specified measure.
  No objective responses were observed. Therefore, duration of response could not be calculated.
Arm/Group | E6201 240 mg/m^2 Weekly | E6201 320 mg/m^2 Weekly | E6201 160 mg/m^2 Twice Weekly | E6201 240 mg/m^2 Twice Weekly | E6201 320 mg/m^2 Twice Weekly
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Progression-Free Survival
Description: Length of time from the date of first administration of study drug to the first evidence of disease progression or death, whichever is earlier
Time Frame: From Cycle 1 Day 1 (C1D1) until death or study closure, up to 26 months
Population: The analysis population was the per-protocol set (PPS). The PPS included all subjects in the FAS who had a valid baseline and one or more post-treatment assessments for a specified measure.
  For AML, MDS and CMML, progression was defined by relevant IWG criteria as failure to achieve at least a PR.
  No responses; PFS could not be calculated.
Arm/Group | E6201 240 mg/m^2 Weekly | E6201 320 mg/m^2 Weekly | E6201 160 mg/m^2 Twice Weekly | E6201 240 mg/m^2 Twice Weekly | E6201 320 mg/m^2 Twice Weekly
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Overall Survival
Description: Length of time from the date of first administration of study drug to the date of death from any cause
Time Frame: From C1D1 until death or study closure, up to 26 months
Population: The analysis population was the per-protocol set (PPS). The PPS included all subjects in the FAS who had a valid baseline and one or more post-treatment assessments for a specified endpoint.
Measure: Median (Standard Deviation); unit: Days
Arm/Group | E6201 240 mg/m^2 Weekly | E6201 320 mg/m^2 Weekly | E6201 160 mg/m^2 Twice Weekly | E6201 240 mg/m^2 Twice Weekly | E6201 320 mg/m^2 Twice Weekly
Number analyzed (Participants) | 3 | 9 | 2 | 2 | 3
Days | 31 (13.01) | 68 (50.39) | 96 (69.30) | 99 (48.08) | 30 (35.37)

7. Secondary Outcome: Pharmacokinetic Profile of E6201 in Plasma: Cmax
Description: Cmax: Maximum measured plasma concentration over the collection period
Time Frame: Assessed at Cycle 1 Days 1 and 15, Cycle 2 Day 1, pre-dose, 5 minutes following the end of the 2-hour infusion, 2, 4, 8 and 24 hours post-infusion. Summary PK parameters for Cycle 1 Day 1 reported.
Population: All subjects in the FAS who completed at least 1 pharmacokinetic (PK) assessment.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | E6201 240 mg/m^2 Weekly | E6201 320 mg/m^2 Weekly | E6201 160 mg/m^2 Twice Weekly | E6201 240 mg/m^2 Twice Weekly | E6201 320 mg/m^2 Twice Weekly
Number analyzed (Participants) | 7 | 10 | 3 | 3 | 4
ng/mL | 1195.04 (10.6) | 1430.39 (76.2) | 736.87 (50.7) | 941.66 (47.7) | 1681.12 (5.6)

8. Secondary Outcome: Pharmacokinetics of E6201 in Plasma: Tmax
Description: Tmax: Time to maximum measured plasma concentration
Time Frame: as for outcome 7
Population: All subjects in the FAS who completed at least 1 pharmacokinetic (PK) assessment.
Measure: Mean (Standard Deviation); unit: h
Groups:
- E6201 240 mg/m^2 Weekly: E6201 240 mg/m^2 administered IV over 2 hours once weekly, on Days 1, 8, 15, and 22, repeated every 28 days (= 1 cycle) until progression of disease, toxicity or other reason for discontinuation of study drug, and followed for up to 6 months after the last dose.
- E6201 320 mg/m^2 Weekly: E6201 320 mg/m^2 administered IV over 2 hours once weekly, on Days 1, 8, 15, and 22, repeated every 28 days (= 1 cycle) until progression of disease, toxicity or other reason for discontinuation of study drug, and followed for up to 6 months after the last dose.
- E6201 160 mg/m^2 Twice Weekly: E6201 160 mg/m^2 administered IV over 2 hours twice weekly, on Days 1, 4, 8, 11, 15, 18, 22 and 25, repeated every 28 days (= 1 cycle) until progression of disease, toxicity or other reason for discontinuation of study drug, and followed for up to 6 months after the last dose.
- E6201 240 mg/m^2 Twice Weekly: E6201 240 mg/m^2 administered IV over 2 hours twice weekly, on Days 1, 4, 8, 11, 15, 18, 22 and 25, repeated every 28 days (= 1 cycle) until progression of disease, toxicity or other reason for discontinuation of study drug, and followed for up to 6 months after the last dose.
- E6201 320 mg/m^2 Twice Weekly: E6201 320 mg/m^2 administered IV over 2 hours twice weekly, on Days 1, 4, 8, 11, 15, 18, 22, and 25, repeated every 28 days (= 1 cycle) until progression of disease, toxicity or other reason for discontinuation of study drug, and followed for up to 6 months after the last dose.
Arm/Group | E6201 240 mg/m^2 Weekly | E6201 320 mg/m^2 Weekly | E6201 160 mg/m^2 Twice Weekly | E6201 240 mg/m^2 Twice Weekly | E6201 320 mg/m^2 Twice Weekly
Number analyzed (Participants) | 7 | 10 | 3 | 3 | 4
h | 2.34 (7.5) | 4.10 (95.4) | 2.17 (0.9) | 2.32 (6.8) | 2.18 (4.2)

9. Secondary Outcome: Pharmacokinetic Profile of E6201 in Plasma: AUCT
Description: Area under the plasma concentration versus time curve (AUC) to the last measurable concentration over the sampling time-interval.
Time Frame: as for outcome 7
Population: All subjects in the FAS who completed at least 1 pharmacokinetic (PK) assessment.
Measure: Mean (Standard Deviation); unit: h.ng/mL
Arm/Group | E6201 240 mg/m^2 Weekly | E6201 320 mg/m^2 Weekly | E6201 160 mg/m^2 Twice Weekly | E6201 240 mg/m^2 Twice Weekly | E6201 320 mg/m^2 Twice Weekly
Number analyzed (Participants) | 7 | 10 | 3 | 3 | 4
h.ng/mL | 3797.76 (20.6) | 8135.24 (88.0) | 3034.10 (69.8) | 2796.73 (50.3) | 6082.79 (23.0)

10. Secondary Outcome: Pharmacokinetic Profile of E6201 in Plasma: AUCI
Description: AUCI: The area under the concentration versus time curve from time 0 to infinity
Time Frame: as for outcome 7
Population: All subjects in the FAS who completed at least 1 pharmacokinetic (PK) assessment.
Measure: Mean (Standard Deviation); unit: h.ng/mL
Arm/Group | E6201 240 mg/m^2 Weekly | E6201 320 mg/m^2 Weekly | E6201 160 mg/m^2 Twice Weekly | E6201 240 mg/m^2 Twice Weekly | E6201 320 mg/m^2 Twice Weekly
Number analyzed (Participants) | 7 | 10 | 3 | 3 | 4
h.ng/mL | 3871.83 (21.7) | 2506.90 (56.0) | 1853.13 (1.1) | 2215.63 (59.0) | 6388.31 (25.0)

11. Secondary Outcome: Pharmacokinetic Profile of E6201 in Plasma: T1/2
Description: T1/2: The apparent first-order elimination half-life
Time Frame: as for outcome 7
Population: All subjects in the FAS who completed at least 1 pharmacokinetic (PK) assessment.
Measure: Mean (Standard Deviation); unit: h
Arm/Group | E6201 240 mg/m^2 Weekly | E6201 320 mg/m^2 Weekly | E6201 160 mg/m^2 Twice Weekly | E6201 240 mg/m^2 Twice Weekly | E6201 320 mg/m^2 Twice Weekly
Number analyzed (Participants) | 7 | 10 | 3 | 3 | 4
h | 3.78 (88.0) | 2.71 (87.5) | 3.20 (43.6) | 1.66 (4.5) | 5.01 (71.1)

12. Secondary Outcome: Pharmacokinetic Profile of E6201 in Plasma: CLobs
Description: Clearance observed (CLobs): Total body clearance for extravascular administration
Time Frame: as for outcome 7
Population: All subjects in the FAS who completed at least 1 pharmacokinetic (PK) assessment.
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | E6201 240 mg/m^2 Weekly | E6201 320 mg/m^2 Weekly | E6201 160 mg/m^2 Twice Weekly | E6201 240 mg/m^2 Twice Weekly | E6201 320 mg/m^2 Twice Weekly
Number analyzed (Participants) | 7 | 10 | 3 | 3 | 4
L/h | 104.0 (17.8) | 300.2 (45.3) | 150.68 (15.3) | 221.2 (70.1) | 85.7 (33.1)

13. Secondary Outcome: Pharmacokinetic Profile of E6201 in Plasma: VDobs
Description: Measurement of apparent volume of distribution observed (VDobs)
Time Frame: as for outcome 7
Population: All subjects in the FAS who completed at least 1 pharmacokinetic (PK) assessment.
Measure: Mean (Standard Deviation); unit: L
Arm/Group | E6201 240 mg/m^2 Weekly | E6201 320 mg/m^2 Weekly | E6201 160 mg/m^2 Twice Weekly | E6201 240 mg/m^2 Twice Weekly | E6201 320 mg/m^2 Twice Weekly
Number analyzed (Participants) | 7 | 10 | 3 | 3 | 4
L | 523.1 (76.2) | 940.6 (52.6) | 718.56 (57.0) | 536.5 (73.4) | 523.6 (42.4)

14. Secondary Outcome: Number of Participants With Suppression of pERK at 4 Hours Post-dose
Description: phospho-ERK (pERK) in blood assessed by Western blot at 4 hours post-dose
Time Frame: Cycle 1 Day 1, 4 hours post-dose.
Population: All subjects in the FAS who completed at least 1 PD assessment. Data obtained were not quantitative.
Measure: Count of Participants; unit: Participants
Arm/Group | E6201 240 mg/m^2 Weekly | E6201 320 mg/m^2 Weekly | E6201 160 mg/m^2 Twice Weekly | E6201 240 mg/m^2 Twice Weekly | E6201 320 mg/m^2 Twice Weekly
Number analyzed (Participants) | 7 | 10 | 3 | 3 | 4
Participants | 3 | 2 | 2 | 2 | 1

15. Secondary Outcome: Number of Participants With Suppression of pERK at 24 Hours Post-dose
Description: Measurement of phospho-ERK (pERK) in blood assessed by Western blot at 24 hours post-dose
Time Frame: Cycle 1 Day 1, 24 hours post-dose.
Population: All subjects in the FAS who completed at least 1 PD assessment. Data obtained were not quantitative.
Measure: Count of Participants; unit: Participants
Arm/Group | E6201 240 mg/m^2 Weekly | E6201 320 mg/m^2 Weekly | E6201 160 mg/m^2 Twice Weekly | E6201 240 mg/m^2 Twice Weekly | E6201 320 mg/m^2 Twice Weekly
Number analyzed (Participants) | 7 | 10 | 3 | 3 | 4
Participants | 2 | 1 | 2 | 1 | 0

16. Secondary Outcome: Number of Participants With Suppression of pFLT3 at 4 Hours Post-dose
Description: phospho-FLT3 (pFLT3) in blood assessed by Western blot at 4 hours post-dose
Time Frame: Cycle 1 Day 1, 4 hours post-dose.
Population: All subjects in the FAS who completed at least 1 PD assessment. Data obtained were not quantitative.
Measure: Count of Participants; unit: Participants
Arm/Group | E6201 240 mg/m^2 Weekly | E6201 320 mg/m^2 Weekly | E6201 160 mg/m^2 Twice Weekly | E6201 240 mg/m^2 Twice Weekly | E6201 320 mg/m^2 Twice Weekly
Number analyzed (Participants) | 7 | 10 | 3 | 3 | 4
Participants | 3 | 1 | 1 | 2 | 0

17. Secondary Outcome: Number of Participants With Suppression of pFLT3 at 24 Hours Post-dose
Description: phospho-FLT3 (pFLT3) in blood assessed by Western blot at 24 hours post-dose
Time Frame: Cycle 1 Day 1, 24 hours post-dose.
Population: All subjects in the FAS who completed at least 1 PD assessment. Data obtained were not quantitative.
Measure: Count of Participants; unit: Participants
Arm/Group | E6201 240 mg/m^2 Weekly | E6201 320 mg/m^2 Weekly | E6201 160 mg/m^2 Twice Weekly | E6201 240 mg/m^2 Twice Weekly | E6201 320 mg/m^2 Twice Weekly
Number analyzed (Participants) | 7 | 10 | 3 | 3 | 4
Participants | 0 | 1 | 1 | 1 | 0

18. Secondary Outcome: Number of Participants With Suppression of pAKT at 4 Hours Post-dose
Description: phospho-AKT (pAKT) in blood assessed by Western blot at 4 hours post-dose
Time Frame: Cycle 1 Day 1, 4 hours post-dose.
Population: All subjects in the FAS who completed at least 1 PD assessment. Data obtained were not quantitative.
Measure: Count of Participants; unit: Participants
Arm/Group | E6201 240 mg/m^2 Weekly | E6201 320 mg/m^2 Weekly | E6201 160 mg/m^2 Twice Weekly | E6201 240 mg/m^2 Twice Weekly | E6201 320 mg/m^2 Twice Weekly
Number analyzed (Participants) | 7 | 10 | 3 | 3 | 4
Participants | 0 | 0 | 0 | 0 | 0

19. Secondary Outcome: Number of Participants With Suppression of pAKT at 24 Hours Post-dose
Description: phospho-AKT (pAKT) in blood assessed by Western blot at 24 hours post-dose
Time Frame: Cycle 1 Day 1, 24 hours post-dose.
Population: All subjects in the FAS who completed at least 1 PD assessment. Data obtained were not quantitative.
Measure: Count of Participants; unit: Participants
Arm/Group | E6201 240 mg/m^2 Weekly | E6201 320 mg/m^2 Weekly | E6201 160 mg/m^2 Twice Weekly | E6201 240 mg/m^2 Twice Weekly | E6201 320 mg/m^2 Twice Weekly
Number analyzed (Participants) | 7 | 10 | 3 | 3 | 4
Participants | 0 | 0 | 0 | 0 | 0

20. Secondary Outcome: Number of Participants With Suppression of pERK by PIA at 4 Hours Post-dose
Description: Blood assay: Plasma inhibitory assay (PIA) measuring pERK in blood at 4 hours post-dose
Time Frame: Cycle 1 Day 1, 4 hours post-dose.
Population: All subjects in the FAS who completed at least 1 PD assessment. Data obtained were not quantitative.
Measure: Count of Participants; unit: Participants
Arm/Group | E6201 240 mg/m^2 Weekly | E6201 320 mg/m^2 Weekly | E6201 160 mg/m^2 Twice Weekly | E6201 240 mg/m^2 Twice Weekly | E6201 320 mg/m^2 Twice Weekly
Number analyzed (Participants) | 7 | 10 | 3 | 3 | 4
Participants | 7 | 5 | 2 | 3 | 2

21. Secondary Outcome: Number of Participants With Suppression of in pERK by PIA 24 Hours Post-dose
Description: Blood assay: Plasma inhibitory assay (PIA) measuring pERK in blood at 24 hours post-dose
Time Frame: Cycle 1 Day 1, 24 hours post-dose.
Population: All subjects in the FAS who completed at least 1 PD assessment. Data obtained were not quantitative.
Measure: Count of Participants; unit: Participants
Arm/Group | E6201 240 mg/m^2 Weekly | E6201 320 mg/m^2 Weekly | E6201 160 mg/m^2 Twice Weekly | E6201 240 mg/m^2 Twice Weekly | E6201 320 mg/m^2 Twice Weekly
Number analyzed (Participants) | 7 | 10 | 3 | 3 | 4
Participants | 1 | 2 | 1 | 0 | 1

22. Secondary Outcome: Number of Participants With Suppression of pFLT3 by PIA at 4 Hours Post-dose
Description: Blood assay: Plasma inhibitory assay (PIA) measuring pFLT3 in blood at 4 hours post-dose
Time Frame: Cycle 1 Day 1, 4 hours post-dose.
Population: All subjects in the FAS who completed at least 1 PD assessment. Data obtained were not quantitative.
Measure: Count of Participants; unit: Participants
Arm/Group | E6201 240 mg/m^2 Weekly | E6201 320 mg/m^2 Weekly | E6201 160 mg/m^2 Twice Weekly | E6201 240 mg/m^2 Twice Weekly | E6201 320 mg/m^2 Twice Weekly
Number analyzed (Participants) | 7 | 10 | 3 | 3 | 4
Participants | 6 | 5 | 2 | 3 | 2

23. Secondary Outcome: Number of Participants With Suppression of pFLT3 by PIA at 24 Hours Post-dose
Description: Blood assay: Plasma inhibitory assay (PIA) measuring pFLT3 in blood at 24 hours post-dose
Time Frame: Cycle 1 Day 1, 24 hours post-dose.
Population: All subjects in the FAS who completed at least 1 PD assessment. Data obtained were not quantitative.
Measure: Count of Participants; unit: Participants
Arm/Group | E6201 240 mg/m^2 Weekly | E6201 320 mg/m^2 Weekly | E6201 160 mg/m^2 Twice Weekly | E6201 240 mg/m^2 Twice Weekly | E6201 320 mg/m^2 Twice Weekly
Number analyzed (Participants) | 7 | 10 | 3 | 3 | 4
Participants | 1 | 2 | 1 | 0 | 1

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for each subject from C1D1 to 6 months after the last dose of study drug. The total duration of the study was 26 months.
Description: Adverse events were reported for all study participants who were administered any fraction of a dose of study medication.
Arm/Group | E6201 240 mg/m^2 Weekly | E6201 320 mg/m^2 Weekly | E6201 160 mg/m^2 Twice Weekly | E6201 240 mg/m^2 Twice Weekly | E6201 320 mg/m^2 Twice Weekly
All-Cause Mortality (participants affected / at risk) | 3/7 | 4/10 | 1/3 | 0/3 | 1/4
Serious Adverse Events (participants affected / at risk) | 4/7 | 10/10 | 3/3 | 2/3 | 2/4
Other Adverse Events (participants affected / at risk) | 7/7 | 10/10 | 3/3 | 3/3 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | E6201 240 mg/m^2 Weekly (N=7) | E6201 320 mg/m^2 Weekly (N=10) | E6201 160 mg/m^2 Twice Weekly (N=3) | E6201 240 mg/m^2 Twice Weekly (N=3) | E6201 320 mg/m^2 Twice Weekly (N=4)
GI hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 | 0 | 0 | 0
Tumor lysis syndrome (Metabolism and nutrition disorders) | 1 (1) | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 (1) | 2 (2) | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 (1) | 0 | 0 | 0 | 0
Multi-organ failure (General disorders) | 1 (1) | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 (1) | 3 (3) | 1 (1) | 1 | 1 (1)
Alpha hemolytic Strep infection (Infections and infestations) | 1 (1) | 0 | 0 | 0 | 0
Pseudomonal bateremia (Infections and infestations) | 0 | 1 (1) | 0 | 0 | 0
ECG QTc prolonged (Investigations) | 0 | 1 (1) | 0 | 0 | 0
Intracranial hemorrhage (Nervous system disorders) | 0 | 2 (2) | 0 | 0 | 0
Klebsiella bacteremia (Infections and infestations) | 0 | 1 (2) | 0 | 0 | 0
Respiratory tract infection fungal (Infections and infestations) | 0 | 1 (1) | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 (1) | 0 | 1 (3) | 0
Pneumonia (Infections and infestations) | 0 | 3 (7) | 0 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (1) | 1 (1) | 0 | 0
Epiglottitis (Infections and infestations) | 0 | 0 | 1 (1) | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 (1) | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 1 (1) | 0 | 0
Perirectal abscess (Infections and infestations) | 0 | 0 | 0 | 1 (1) | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 (1) | 0
Lobar pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 (1)
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | E6201 240 mg/m^2 Weekly (N=7) | E6201 320 mg/m^2 Weekly (N=10) | E6201 160 mg/m^2 Twice Weekly (N=3) | E6201 240 mg/m^2 Twice Weekly (N=3) | E6201 320 mg/m^2 Twice Weekly (N=4)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 3 | 0 | 2 | 1
Leucocytosis (Blood and lymphatic system disorders) | 1 | 3 | 0 | 1 | 0
Spleen disorder (Blood and lymphatic system disorders) | 1 | 2 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 0 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 2 | 1 | 0 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 1
Nausea (Gastrointestinal disorders) | 2 | 2 | 0 | 1 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 2 | 0 | 1 | 0
Chills (General disorders) | 0 | 0 | 1 | 1 | 0
Fatigue (General disorders) | 1 | 2 | 1 | 1 | 2
Non-cardiac chest pain (General disorders) | 0 | 1 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 2 | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 1 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 3 | 0 | 0 | 0
Pneumonia fungal (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 | 3 | 1 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 2 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 2 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 0 | 0
ALT increased (Investigations) | 1 | 0 | 1 | 2 | 0
AST increased (Investigations) | 1 | 0 | 1 | 1 | 1
ECG QT prolonged (Investigations) | 1 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 2 | 0 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1
Fluid overload (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 1 | 1
Hemorrhage intracranial (Nervous system disorders) | 0 | 2 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 2 | 1 | 0 | 1
Mental disorder (Psychiatric disorders) | 2 | 0 | 0 | 0 | 0
Hematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 2 | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 2 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 1
Pruritis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 2 | 1 | 1 | 0

LIMITATIONS AND CAVEATS:
Although E6201 exhibited an acceptable safety profile when administered at doses up to the MTD of 320 mg/m^2 IV twice weekly, insufficient efficacy was observed during the Phase 1 portion of the study. Thus, the Phase 2a portion was not initiated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-10-19): https://cdn.clinicaltrials.gov/large-docs/00/NCT02418000/SAP_000.pdf
  • Study Protocol (2016-10-30): https://cdn.clinicaltrials.gov/large-docs/00/NCT02418000/Prot_001.pdf